CLINICAL TRIAL: NCT01372644
Title: Breast Cancer Chemoprevention by SOM230, an IGF-I Action Inhibitor: A Proof of Principle Trial
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R6-937; BC061512 (Other Grant/Funding Number: Department of Defense)
Record Dates: First submitted 2011-06-09; First posted 2011-06-14 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-12

CONDITIONS: Atypical Ductal Breast Hyperplasia; Lobular Carcinoma in Situ (LCIS); Atypical Lobular Hyperplasia (ALH) of Breast
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating; Breast Carcinoma In Situ | interventions — pasireotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ADH, ALH, LCIS, SOM 230 (Experimental): Women who meet eligibility criteria.
  Interventions: Drug: SOM 230 / Pasireotide

INTERVENTIONS:
Drug: SOM 230 / Pasireotide

SUMMARY:
Atypical ductal hyperplasia (ADH) and atypical lobular hyperplasia (ALH) increases breast cancer risk. In post menopausal women, SERMS are standard chemopreventive agents. The investigators have previously shown insulin-like growth factor-I (IGF-I) is required to permit estrogen (E2) and progesterone action in the mammary gland, and that a novel somatostatin analog, SOM230, that inhibits IGF-I action can prevent E2 action on the mammary gland. It reduces cell proliferation and increases apoptosis (cell death) in the rat mammary gland. This study was designed to determine whether women at high risk for breast cancer respond to SOM230 in the same way that rats do. Methods: Women with atypical ductal hyperplasia or lobular carcinoma in-situ by core biopsy were treated for 9.5 days with SOM230 (600mcg BID). Surgical excision was performed on day 10. Sections were examined before and after SOM230 treatment for cell proliferation (Ki67) and apoptosis (TUNEL). Serum IGF-I, fasting glucose, insulin, and HbA1C were measured in anticipation of changes.

ELIGIBILITY:
Inclusion Criteria

* Over 21 years of age
* Must sign informed consent, witnessed, and dated prior to entry
* The participant has an increased risk for developing breast cancer which may include; Atypical Ductal Hyperplasia (ADH), Lobular Carcinoma in situ (LCIS), and/or Atypical Lobular Hyperplasia (ALH)
* Performance Status: ECOG 0-1 unless mobility is limited from chronic physical handicap
* No clinical evidence of other malignancies (except Basal Cell carcinoma)
* Complete blood count, differential and platelet count must be within normal limits (WNL) or verified by the study chair to be related to conditions not interfering with normal health status
* Adequate hepatic and renal function (these must be WNL or verified by study chair to be related to conditions not interfering with normal health status)
* Normal fasting glucose
* No history of diabetes
* Medically and Psychologically able to comply with all study requirements
* Accessible to Follow up

Exclusion Criteria

* Less than 21 years of age
* Known invasive breast cancer of any type
* Bilateral prophylactic mastectomy
* Prior malignancy of any type that occurred less than 5 years previously, except for basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix
* Existing non-malignant disease that would preclude the administration of SOM230
* Pregnancy: All subjects will have a beta human chorionic gonadotropin (b-hCG) serum pregnancy test to rule out pregnancy, a history will also be taken to make certain that recent sexual exposure does not put them at risk for pregnancy. If so a second serum pregnancy test will be done. Volunteers will be asked to use barrier contraception during study.
* Tamoxifen or other preventive measures within 6 months
* Serious Psychiatric condition or addictive disorder
* Diabetes or elevated fasting blood sugar
* Inability to inject medication or test for finger stick glucose
* Symptomatic gallstones or known gall bladder disease
* History of cholecystitis without cholecystectomy
* Electrolyte abnormalities (particularly hypokalemia or hypomagnesemia)

QT related exclusion criteria

* QTcF at screening > 450 msec.
* History of syncope or family history of idiopathic sudden death.
* Sustained or clinically significant cardiac arrhythmias.
* Risk factors for Torsades de Pointes such as hypokalemia, hypomagnesemia, cardiac failure, clinically significant/symptomatic bradycardia, or high-grade AV block.
* Concomitant disease(s) that could prolong QT such as autonomic neuropathy (caused by diabetes, or Parkinson's disease), HIV, cirrhosis, uncontrolled hypothyroidism or cardiac failure
* Concomitant medication(s) known to increase the QT interval.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-11; Primary Completion 2010-12 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Cell Proliferation and apoptosis | 10 days
  Tissue from initial diagnostic breast biopsies will be compared to the remaining tissue excised after treatment with SOM230. Tissue will be stained to measure cell proliferation and apoptosis (cell death).

CONTACTS AND LOCATIONS:
Overall Officials: David L Kleinberg, MD, Principal Investigator — NYU School of Medicine; Julia Smith, MD, Study Director — NYU School of Medicine; Deborah Axelrod, MD, Study Director — NYU School of Medicine
Locations (1):
- NYU School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Singh B, Smith JA, Axelrod DM, Ameri P, Levitt H, Danoff A, Lesser M, de Angelis C, Illa-Bochaca I, Lubitz S, Huberman D, Darvishian F, Kleinberg DL. Insulin-like growth factor-I inhibition with pasireotide decreases cell proliferation and increases apoptosis in pre-malignant lesions of the breast: a phase 1 proof of principle trial. Breast Cancer Res. 2014 Nov 11;16(6):463. doi: 10.1186/s13058-014-0463-1. PMID 25385439